CLINICAL TRIAL: NCT03837938
Title: Multicenter Open-label Randomized Clinical Trial of the Efficacy and Safety of Levopront® Syrup 30 mg/5 ml in Comparison With Libexin® 100 mg Tablets in Patients With Dry Non-productive Cough Caused by Acute Upper Respiratory Infection
Brief Title: Clinical Trial of Efficacy and Safety of Levopront® 30 mg/5 ml in Patients With Dry Cough
Acronym: LDP0114
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDP0114
Record Dates: First submitted 2019-01-28; First posted 2019-02-12 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-10

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — dipropizine; libexin

STUDY DESIGN:
Masking Description: It is an open-label clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levopront® syrup 30 mg/5 ml (Experimental): Levopront® (levodropropizine) syrup 30 mg/5 ml 10 ml (60 mg) t.i.d. for 7 days. The study drugs was taken 3 times a day, at intervals of at least 6 hours, between meals for 7 days.
  Interventions: Drug: Levopront® syrup 30 mg/5 ml
- Libexin® 100 mg tablets (Active Comparator): Libexin® (prenoxdiazine) 100 mg tablets. Libexin® was administered orally, 1 tablet (100 mg) 3 times a day for 7 days.
  Interventions: Drug: Libexin®

INTERVENTIONS:
Drug: Levopront® syrup 30 mg/5 ml — The first study drug administration was performed at the clinical site on the day of randomization; the last study drug administration was performed in the evening before Day 8 (±1).
  Other Names: levodropropizine
  Arms: Levopront® syrup 30 mg/5 ml
Drug: Libexin® — The first study drug administration was performed at the clinical site on the day of randomization; the last study drug administration was performed in the evening before Day 8 (±1). No chewing.
  Other Names: prenoxdiazine
  Arms: Libexin® 100 mg tablets

SUMMARY:
Primary objective:

To assess the efficacy of Levopront® in comparison with Libexin® based on daytime cough resolution rate by Day 8.

The daytime cough symptoms resolution corresponds to 0 or 1 points on the "Six-point daytime and nighttime cough assessment scale".

Secondary objectives:

Treatment effect assessment in terms of the following efficacy and safety parameters:

* To assess the efficacy of Levopront® in comparison with Libexin® based on nighttime cough resolution rate by Day 8.
* Daytime and nighttime cough symptoms resolution according to "Six-point daytime and nighttime cough assessment scale" by Day 4.
* Change in severity and frequency of daytime and nighttime cough according to "Six-point daytime and nighttime cough assessment scale" on Day 4 and Day 8 from baseline on Day 1.
* Cough intensity change according to the visual-analogue scale on Day 4 and Day 8 from baseline on Day 1.
* Change of FEV1 on Day 8 from baseline values on Day 1.
* Rate of Adverse events (AE) and Serious Adverse Events (SAE) of the various severity according to subjective complaints, laboratory test results, physical examination, vital signs and spirometry

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, clinical trial to assess the efficacy and safety of Levopront® syrup 30 mg/5 ml in comparison with Libexin® 100 mg tablets in patients suffering from dry non-productive cough caused by acute upper respiratory infection

ELIGIBILITY:
Inclusion Criteria:

Subjects should meet the following inclusion criteria to be included into this clinical trial:

1. Signed Informed Consent Form
2. Male or female aged from 18 to 65 (inclusive)
3. Dry non-productive cough as a symptom of acute upper respiratory infection (IDC codes J00-J06)
4. Daytime cough symptom score ≥ 3 points according to the "Six-point daytime and nighttime cough assessment scale"
5. Pre-bronchodilator FEV1 ≥ 70% of the predicted values, post-bronchodilator FEV1 increase of ≤ 12% or ≤ 200 ml compared to the baseline, FEV1/FVC (Tiffeneau index) ≥ 0.7
6. Patient's consent to follow the protocol procedures, including the completion of the patient's diary
7. Patient's consent to use the adequate contraception methods throughout the study period. The adequate birth control methods are as follows:

   * Oral or transdermal contraceptives
   * Condoms or diaphragms (barrier method) with spermicide
   * Intrauterine contraceptive devices

Exclusion Criteria:

Subjects with any of the following conditions will be excluded from the study:

1. Hypersensitivity or individual contraindications to Levodropropizine, Prenoxdiazine or additives of the study drug
2. Hereditary fructose intolerance, glucose-lactose malabsorption, lactase deficiency, sucrose-isomaltose deficiency
3. Tuberculosis, bronchial asthma, malignant tumors of lungs or bronchi, COPD, severe respiratory failure (cyanosis, need for respiratory support) or other lung pathology at screening or in history
4. Inhalation anesthesia within 3 months before screening
5. Smoking history of more than 10 pack-years
6. Previous use of cough medicines, ACE inhibitors or amiodarone within 30 days before screening
7. Contraindications or inability to perform spirometry
8. Necessity (in the Investigator's opinion) of prescribing mucolytic agents, expectorants, antibiotics or other medications prohibited by the protocol during the study
9. Excessive mucous excretion which (in the Investigator's opinion) could be a contraindication to prescribing anti-cough medicines; decreased mucociliary function (Kartagener's syndrome, ciliary dyskinesia)
10. Malignant tumors in the past 5 years (except for the basal cell carcinoma)
11. Serious cardiovascular disease at the moment or within 12 months prior to screening, including: Chronic heart failure class III or IV (according to the classification of the New York Heart Association), severe arrhythmias requiring treatment with antiarrhythmic drugs class Ia, Ib, Ic or III, unstable angina, myocardial infarction, heart surgery and coronary arteries, serious valvular heart disease, transient ischemic attack or stroke, uncontrolled hypertension with systolic blood pressure > 180 mmHg and diastolic blood pressure > 110 mmHg, pulmonary embolism or deep vein thrombosis
12. Gastric or duodenal ulcers, gastroesophageal reflux disease within a period of 12 months before screening
13. Systemic autoimmune disorders and connective tissue diseases that require (currently or previously) administration of systemic glucocorticosteroids, cytostatic medications or penicillamine
14. Signs of intensive non-controlled concurrent disease, including disorders of the nervous system, endocrine system, kidneys, liver or gastrointestinal tract, which (in the Investigator's opinion) could prevent the patient's participation in the study
15. History of alcohol or drug abuse at screening or in the past, which results in the inability of the patient to participate in the study at the Investigator's discretion
16. Taking part in another clinical trial or use of study drug within 30 days before screening
17. Pregnant or breast-feeding women or women planning pregnancy during the clinical trial; women of childbearing potential (including not sterilized operatively and in postmenopausal period of less than 2 years), not using appropriate methods of contraception
18. Inability to read or write; unwillingness to understand and follow the procedures of the study protocol; violation of the drug administration regimen or procedure execution that, at the discretion of the Investigator, can impact he results of the study or safety of the patient and interfere his further participation in the study; any other concomitant medical or serious mental conditions that make the patient unsuitable for participation in the clinical study, limit the validity of receiving an informed consent or may affect the patient's ability to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Saibene, MD, Study Director — Dompé SpA Milan
Locations (8):
- Russia (8):
  - State Public Healthcare Institution of Moscow "City Clinical Hospital # 71 of Moscow Healthcare Department", Moscow
  - The Laboratory of Pulmonology, State Budgetary Educational Institution of Higher Professional Education "Moscow State Medical-Stomatological University n.a. A.I. Evdokimov" under Ministry of Health of the Russian Federation (Clinical base of state budget, Moscow
  - State Budgetary Educational Institution of Higher Professional Education "Ryazan' State Medical University n.a. academician I.P. Pavlov" under Ministry of Health of the Russian Federation, Ryazan
  - "Institute of Medical Research" LLC, Saint Petersburg
  - Saint-Petersburg State Healthcare Institution "Nikolaevskaya Hospital", Saint Petersburg
  - State Healthcare Institution "Regional Clinical Hospital", Saratov
  - LLC Treatment-and-prophylactic institution on the "Smolensk clinic", Smolensk
  - State Autonomous Healthcare Institution of Yaroslavl Region "Clinical Hospital of Emergency care n.a. N.V. Solovyev", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Totally, 184 patients were randomized into Levopront® (Test) and the Libexin® (Control) treatment groups: there were 92 patients in each group. All the patients completed the study according to the protocol. One patient was screen failure due to post-bronchodilator FEV1 increase.
Period: Overall Study
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets
Started | 92 | 92
ITT Population | 92 | 92
PP Population | 88 | 91
Safety Population | 92 | 92
Completed | 92 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT population consisted of all randomized patients from both treatment groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92 | 92 | 184
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (11.4) | 40.2 (13.4) | 40.2 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 64 | 124
  Male | 32 | 28 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 92 | 92 | 184
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 92 | 92 | 184

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Daytime Cough Resolution Rate by Day 8 in the PP Population
Description: Daytime cough (>08:00h up to 22:00 h) was evaluated on a 6-point scale (Six-point daytime and nighttime cough assessment scale") where 0 = no cough during the day; and 5 = distressing cough most of the day. The daytime cough symptoms resolution corresponds to 0 or 1 points on the 6-point scale. The lower the score the better the outcome.
  The rate of patients who responded to treatment (cough absents, when score is 0 or 1 at "six-point cough scale" vs. cough presents, when score is ≥ 2 at "six-point cough score") by Day 8 in the study treatment group and in the control group with a non-inferiority margin of δ = 20% is reported.
Time Frame: At Visit 3, Day 8
Population: Per-Protocol population included all randomized patients completing treatment with the study drug, having primary efficacy analysis assessment done and considered to be compliant.
Measure: Count of Participants; unit: Participants
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets
Number analyzed (Participants) | 88 | 91
Participants
  Resolved (<2) | 67 | 64
  Ongoing (≥2) | 21 | 27
Statistical Analysis 1: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; Difference in daytime resolved rates Levopront® (Test) vs Libexin® (Control) was reported; Test type: Non-Inferiority — According to the protocol and SAP non-inferiority margin was defined as 20%; Difference in rates Levopront®-Libexin® = 5.81, 97.5% CI 1-sided [lower limit -7.17]

2. Primary Outcome: Number of Participants With Daytime Cough Resolution Rate by Day 8 in the ITT Population
Description: as for outcome 1
Time Frame: At Visit 3, Day 8
Population: ITT population: the population of patients based on the initial treatment assignment and not on the treatment eventually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets
Number analyzed (Participants) | 92 | 92
Participants
  Resolved (<2) | 70 | 65
  Ongoing (≥2) | 22 | 27
Statistical Analysis 1: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; Difference in daytime resolved rates Levopront® (Test) vs Libexin® (Control) was reported; Test type: Non-Inferiority — According to the protocol and SAP non-inferiority margin was defined as 20%; difference in rates Levopront®-Libexin® = 5.43, 97.5% CI 1-sided [lower limit -7.31]

3. Secondary Outcome: Number of Participants With Nighttime Cough Resolution Rate by Day 8 in the ITT Population
Description: Night-time cough ( >22:00 h up to 08:00 h) was evaluated on a 6-point scale (Six-point daytime and nighttime cough assessment scale") where 0 = no cough during the night to 5 = distressing coughs preventing any sleep. The nighttime cough symptoms resolution corresponds to 0 or 1 points on the 6-point scale. The lower the score the better the outcome.
  The rate of patients who responded to treatment (cough absents, when score is 0 or 1 at "six-point cough scale" vs. cough presents, when score is ≥ 2 at "six-point cough score") by Day 8 in the study treatment group and in the control group with a non-inferiority margin of δ = 20% is reported.
Time Frame: At Visit 3, Day 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets
Number analyzed (Participants) | 92 | 92
Participants
  Resolved (<2) | 90 | 89
  Ongoing (≥2) | 2 | 3
Statistical Analysis 1: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; Test type: Non-Inferiority — non-inferiority margin was defined as 20%; p > 0.999, Fisher Exact

4. Secondary Outcome: Number of Participants With Daytime & Nighttime Cough Symptoms Resolution in the ITT Population
Description: Daytime cough ( >08:00h up to 22:00 h) was evaluated on a 6-point scale (Six-point daytime and nighttime cough assessment scale) where 0 = no cough during the day to 5 = distressing coughs most of the day. Night-time cough ( >22:00 h up to 08:00 h) was evaluated on a 6-point scale (Six-point daytime and nighttime cough assessment scale) where 0 = no cough during the night to 5 = distressing coughs preventing any sleep.
  The (daytime and nighttime) cough symptoms resolution corresponds to 0 or 1 points on the 6-point scale. The lower the score the better the outcome.
  The rate of patients who responded to treatment (cough absents, when score is 0 or 1 at "six-point cough scale" vs. cough presents, when score is ≥ 2 at "six-point cough score") by Day 4 in the study treatment group and in the control group with a non-inferiority margin of δ = 20% is reported.
Time Frame: At Visit 2, Day 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets
Number analyzed (Participants) | 92 | 92
Participants
  Resolved (<2) | 22 | 20
  Ongoing (≥2) | 70 | 72
Statistical Analysis 1: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; Test type: Non-Inferiority — non-inferiority margin was defined as 20%; p = 0.861, Fisher Exact

5. Secondary Outcome: Change From Baseline in Severity and Frequency of Daytime and Nighttime Cough According to "Six-point Daytime and Nighttime Cough Assessment Scale" in the ITT Population
Description: Daytime cough ( >08:00 h up to 22:00 h) evaluated on a 6-point scale: 0 = no cough during the day to 5 = distressing coughs most of the day.
  Night-time cough ( >22:00 h up to 08:00 h) evaluated on a 6-point scale: 0 = no cough during the night to 5 = distressing coughs preventing any sleep.
Time Frame: Baseline, At visit 2 Day 4; at visit 3, Day 8
Population: ITT population: the population of patients is based on the initial treatment assignment and not on the treatment eventually received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets
Number analyzed (Participants) | 92 | 92
units on a scale
  daytime cough score at Visit 2, Day 4 | -1.2 (0.8) | -1.2 (0.6)
  daytime cough score at Visit 3, Day 8 | -2.5 (0.8) | -2.2 (0.7)
  nighttime cough score at Visit 2, Day 4 | -0.9 (0.8) | -1.0 (0.9)
  nighttime cough score at Visit 3, Day 8 | -1.9 (1.1) | -1.9 (1.0)
Statistical Analysis 1: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; Daytime at Visit 2, Day 4; Test type: Non-Inferiority — non-inferiority margin was defined as 20%; p < 0.001, t-test, 1 sided; Between groups change was tested using two sample t-test (normal data) or Mann-Whitney test (violation of normality)
Statistical Analysis 2: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; Daytime at Visit 3, Day 8; Test type: Non-Inferiority — non-inferiority margin was defined as 20%; p < 0.001, t-test, 2 sided; Between groups change was tested using two sample t-test (normal data) or Mann-Whitney test (violation of normality)
Statistical Analysis 3: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; Nightime at Visit 2, Day 4; Test type: Non-Inferiority — non-inferiority margin was defined as 20%; p < 0.001, t-test, 1 sided; Between groups change was tested using two sample t-test (normal data) or Mann-Whitney test (violation of normality)
Statistical Analysis 4: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; Nighttime at Visit 3, Day 8; Test type: Non-Inferiority — non-inferiority margin was defined as 20%; p < 0.001, t-test, 1 sided; Between groups change was tested using two sample t-test (normal data) or Mann-Whitney test (violation of normality)

6. Secondary Outcome: Change From Baseline in Cough Intensity According to the Visual-analogue Scale (VAS) in the ITT Population.
Description: The visual-analogue scale (VAS) is a 100 mm scale which ranges from 'no cough' (0 mm) to 'the worst cough severity' (100 mm). The higher the score, the worse the outcome.
Time Frame: Baseline, At visit 2 (Day 4); at visit 3 (Day 8)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets
Number analyzed (Participants) | 92 | 92
units on a scale
  Visit 2, Day 4 | -28.9 (15.0) | -24.9 (15.0)
  Visit 3, Day 8 | -52.1 (18.1) | -44.6 (17.8)
Statistical Analysis 1: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; Visit 2, Day 4; Test type: Non-Inferiority — non-inferiority margin was defined as 20%; p < 0.001, t-test, 1 sided; Between groups change was tested using two sample t-test (normal data) or Mann-Whitney test (violation of normality)
Statistical Analysis 2: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; at Visit 3, Day 8; Test type: Non-Inferiority — non-inferiority margin was defined as 20%; p < 0.001, t-test, 1 sided; Between groups change was tested using two sample t-test (normal data) or Mann-Whitney test (violation of normality)

7. Secondary Outcome: Change From Baseline in Pre-bronchodilator FEV1 Values on Day 8 in the ITT Population.
Description: FEV1 is the Forced Expiratory Volume (in liters) in 1 second. The higher the value, the better the outcome.
Time Frame: At Visit 3 (Day 8)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets
Number analyzed (Participants) | 92 | 92
liters | 0.0 (0.6) | 0.1 (0.4)
Statistical Analysis 1: Comparison: Levopront® Syrup 30 mg/5 ml vs Libexin® 100 mg Tablets; Test type: Non-Inferiority — non-inferiority margin is defined as 20%; p = 0.336, t-test, 1 sided; Between groups change was tested using two sample t-test (normal data) or Mann-Whitney test (violation of normality)

8. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE) of the Various Severity According to Subjective Complaints
Description: Adverse Event (AE) - any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, complaint or disorder.
  Serious Adverse Event (SAE) - Any adverse medical event which, irrespective of the dose of the study drug:
  * results in death;
  * is life-threatening;
  * requires hospitalization (initial or prolonged);
  * results in significant, persistent or permanent impairment or disability; or
  * is a congenital anomaly or birth defect
  * is an important medical event that may be not immediately life threatening or result in death or hospitalization but, based upon appropriate medical judgment, may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in the definition above.
Time Frame: From the moment of signing Informed Consent Form (prior to administration of the first dose of the study drug) to Day 30 after the last visit of the patient or last procedure per protocol, up to day 10"
Population: Safety population: all patients who received at least one dose of the study drug will be included into the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets
Number analyzed (Participants) | 92 | 92
Participants
  patients with AE/SAE | 14 | 12
  patients with SAE | 0 | 0
  Patients with death outcome AE/SAE | 0 | 0
  Patients with mild and moderate AE/SAE | 14 | 12
  Patients with severe AE/SAE | 0 | 0
  Patients with related (possible, probable or highly probable) AE/SAE | 1 | 2
  Patients with AE/SAE led to discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: At visits 1 (day 1), 2 (day 4), 3 (Day 8) and follow-up (telephon call), up to day 10
Arm/Group | Levopront® Syrup 30 mg/5 ml | Libexin® 100 mg Tablets
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/92
Other Adverse Events (participants affected / at risk) | 14/92 | 12/92
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levopront® Syrup 30 mg/5 ml (N=92) | Libexin® 100 mg Tablets (N=92)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 4 (4)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminitransferase increased (Investigations) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Sleep disorders (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT03837938/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03837938/SAP_001.pdf